CLINICAL TRIAL: NCT01803490
Title: Bacterial Colonization of Suction Drains Following Spine Surgery
Status: Completed | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Nimrod Rahamimov, Head of Spine Surgery Unit, Western Galilee Hospital-Nahariya
Other Study IDs: 0076-12-NHR
Record Dates: First submitted 2013-01-23; First posted 2013-03-04 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Surgical Site Infection, Closed Suction Drains
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Closed suction drains are commonly used following surgery, if the wound is expected to discharge significant amounts of fluid. To this date, no evidence base exists as to the exact post operative time period or discharge volume necessitating presence of a drain. In orthopedic common practice, drains are removed on the second post operative day, fearing the drain will serve as a point of entry for nosocomial infection. In this study, drains will be left in place as long as daily discharge volume exceeds 50cc, regardless of the amount of days following surgery. Daily cultures and antibiotic levels will be taken from the drains receptacle, to determine if and when the drains is colonized by aerobic bacteria.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing spine surgery that requires suction draining,and do not meet the exclusion criteria for this study.

Exclusion Criteria:

* Known active infection in the spine or elsewhere.

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing elective or emergent spine surgery in the normal course of activity at the Western Galilee Hospital spine surgery unit.
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2013-01; Primary Completion 2019-04-27 (Actual); Study Completion 2019-04-27 (Actual)

PRIMARY OUTCOMES:
Growth of bacteria in drain fluids | up to 10 days per patient, (from first post operative day until removal of drains).

SECONDARY OUTCOMES:
antibiotic level in drain fluid | up to 10 days per patient (from first post operative day until removal of drains).

CONTACTS AND LOCATIONS:
Overall Officials: nimrod t Rahamimov, md, Principal Investigator — Head, Dept. of Orthopedics and spine surgery
Locations (1):
- Western Galilee Hospital, Nahariya, Israel